CLINICAL TRIAL: NCT01886378
Title: An Open-label Phase 2 Study to Assess Safety and Clinical Effects of UX007 in Subjects With Long-Chain Fatty Acid Oxidation Disorders (LC-FAOD)
Brief Title: A Study of UX007 (Triheptanoin) in Participants With Long-Chain Fatty Acid Oxidation Disorders (LC-FAOD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UX007-CL201; 2013-004830-14 (EudraCT Number)
Expanded Access: NCT03773770 (Available)
Record Dates: First submitted 2013-06-18; First posted 2013-06-25 (Estimated); Results first posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Long-chain Fatty Acid Oxidation Disorders (LC-FAOD); Carnitine Palmitoyltransferase (CPT II) Deficiency; Very Long Chain Acyl-CoA Dehydrogenase (VLCAD) Deficiency; Longchain 3-hydroxy-acyl-CoA Dehydrogenase (LCHAD) Deficiency; Trifunctional Protein (TFP) Deficiency
Keywords: FAOD; VLCAD; CPT II; CPT2; CPT 2; LCHAD; UX007; Triheptanoin; TFP; C7
MeSH Terms: conditions — VLCAD deficiency | interventions — triheptanoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- UX007 (Experimental): UX007 dosing titrated to a target dose of 25-35% of total caloric intake or maximum tolerated dose. Participants are followed to evaluate the effects of UX007 over 24 weeks (Treatment Period), then continued treatment in the Extension Period for an additional 54 weeks for a total of 78 weeks of treatment.
  Interventions: Drug: UX007

INTERVENTIONS:
Drug: UX007
  Other Names: triheptanoin; C7 oil

SUMMARY:
The primary objective of the study was to evaluate the impact of UX007 on acute clinical pathophysiology associated with LC-FAOD following 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CPT II, VLCAD, LCHAD, or TFP deficiency, based on results of acylcarnitine profiles, fatty acid oxidation probe studies in cultured fibroblasts, and/or mutation analysis obtained from medical records.
* Male or female, at least 6 months of age
* Willing and able to complete all aspects of the study through the end of the study. If a minor, have a caregiver(s) willing and able to assist in all applicable study requirements.
* Provide written informed consent (subjects aged ≥ 18 years), or provide written assent (where appropriate) and have a legally authorized representative willing and able to provide written informed consent
* Willing and able to provide access to medical records charting the last 18-24 months of care prior to the study initiation, or from birth for those subjects less than 18 months of age
* No history of serious adverse reactions or known hypersensitivity to triheptanoin
* Currently managed on a stable treatment regimen (including diet), which may include low-fat/high-carbohydrate diet, avoidance of fasting, carnitine and/or medium-chain triglyceride (MCT) oil. The treatment regimen (including diet) should be stable for the last 60 days to assure that changes in the subject's condition are not confounded by recent changes in the treatment regimen that could affect the 4 week run-in evaluation period. Once study drug treatment has started, must be willing to maintain all aspects of the subject's treatment regimen and diet unchanged, other than discontinuation of MCT oil, in order to avoid potential variability of response due to variations in dietary intake.
* Have severe LC-FAOD, as evidenced by ANY ONE of the following significant clinical manifestations despite therapy:

  * Chronic Elevated Creatine Kinase (CK) with Major Clinical Events: Elevated mean CK levels over the last 6 months -1 year (defined as ≥ 2X upper limit of age/gender-matched normal, or ≥ 500 units/L if age-matched reference not established) not associated with an acute rhabdomyolysis event, AND at least two major clinical events (as defined in the protocol) in the last year, or at least four major clinical events over the last two years,
  * Episodic Elevated CK with Reported Muscle Dysfunction: Episodes of elevated CK levels over the last 6 months -1 year (defined as ≥ 2X upper limit of age/gender-matched normal, or ≥ 500 units/L if age-matched reference is not established) not associated with an acute rhabdomyolysis event, AND patient report of frequent muscle fatigue, exercise intolerance, or limitation of exercise,
  * Highly Elevated CK but Asymptomatic: More seriously elevated mean CK levels (defined as ≥ 4X upper limit of age/gender-matched normal, or ≥ 1000 units/L if age-matched reference is not established) consistent with substantial chronic muscle rupture over the last 6 months-1 year, regardless of frequency of hospitalizations or ER events,
  * Frequent Severe Major Medical Episodes (at least 3 within the past year, or 5 within 2 years) of hypoglycemia, rhabdomyolysis, or exacerbation of cardiomyopathy [CM], requiring emergency room [ER]/acute care visits or hospitalizations,
  * Severe Susceptibility to Hypoglycemia (serum glucose <60 mg/dL) after short periods of fasting (less than 4-12 hours, depending on age), with at least 2 events in the last year that require ongoing prophylactic management, OR recurrent symptomatic hypoglycemia (blood glucose levels or clinical symptoms of hypoglycemia) at home requiring intervention ≥ 2 times per week,
  * Evidence of Functional Cardiomyopathy (with echocardiogram (ECHO) within past 90 days documenting poor ejection fraction [EF]) requiring ongoing medical management
* Females who have reached menarche must have a negative pregnancy test at Screening. If sexually active, subject must be willing to use acceptable method of contraception and have additional pregnancy tests during the study.

Exclusion Criteria:

* Diagnosis of carnitine-acylcarnitine translocase (CACT) or CPT I
* Diagnosis of medium-chain acyl-CoA dehydrogenase (MCAD) deficiency, short- or medium-chain FAOD, ketone body metabolism defect, propionic acidemia or methylmalonic acidemia
* Enrolled in a clinical study involving concurrent use of an investigational drug product within the last 30 days, or unwilling to discontinue use of a prohibited medication or other substance that may confound study objectives
* Unwilling to sign informed consent or release of medical records
* Have any co-morbid conditions, including unstable major organ-system disease(s) that in the opinion of the Investigator, places the subject at increased risk of complications, interferes with study participation or compliance, or confounds study objectives

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-02-06 (Actual); Primary Completion 2016-08-25 (Actual); Study Completion 2016-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical
Locations (10):
- United States (7):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Southern Florida, Tampa, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt Medical Center, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah
- United Kingdom (3):
  - Birmingham Children's Hospital, Birmingham
  - National Hospital for Neurology and Neurosurgery, London
  - Great Ormond Street Hospital, London

REFERENCES:
- [Result] Vockley J, Burton B, Berry GT, Longo N, Phillips J, Sanchez-Valle A, Tanpaiboon P, Grunewald S, Murphy E, Humphrey R, Mayhew J, Bowden A, Zhang L, Cataldo J, Marsden DL, Kakkis E. UX007 for the treatment of long chain-fatty acid oxidation disorders: Safety and efficacy in children and adults following 24weeks of treatment. Mol Genet Metab. 2017 Apr;120(4):370-377. doi: 10.1016/j.ymgme.2017.02.005. Epub 2017 Feb 7. PMID 28189603
- [Result] Vockley J, Burton B, Berry GT, Longo N, Phillips J, Sanchez-Valle A, Tanpaiboon P, Grunewald S, Murphy E, Bowden A, Chen W, Chen CY, Cataldo J, Marsden D, Kakkis E. Results from a 78-week, single-arm, open-label phase 2 study to evaluate UX007 in pediatric and adult patients with severe long-chain fatty acid oxidation disorders (LC-FAOD). J Inherit Metab Dis. 2019 Jan;42(1):169-177. doi: 10.1002/jimd.12038. PMID 30740733
- [Derived] Vockley J, Burton BK, Berry G, Longo N, Phillips J, Sanchez-Valle A, Chapman KA, Tanpaiboon P, Grunewald S, Murphy E, Lu X, Rahman S, Ray K, Reineking B, Pisani L, Ramirez AN. Triheptanoin for the treatment of long-chain fatty acid oxidation disorders: Final results of an open-label, long-term extension study. J Inherit Metab Dis. 2023 Sep;46(5):943-955. doi: 10.1002/jimd.12640. Epub 2023 Jun 19. PMID 37276053
- [Derived] Vockley J, Longo N, Madden M, Dwyer L, Mu Y, Chen CY, Cataldo J. Dietary management and major clinical events in patients with long-chain fatty acid oxidation disorders enrolled in a phase 2 triheptanoin study. Clin Nutr ESPEN. 2021 Feb;41:293-298. doi: 10.1016/j.clnesp.2020.11.018. Epub 2020 Dec 25. PMID 33487279

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following the signing of informed consent at the Screening visit, each participant continued on current long-chain fatty acid oxidation disorder (LC-FAOD) management for a 4-week Run-in Period to establish a clinical baseline. Following completion of the 4-week Run-in Period, participants discontinued any use of medium chain triglycerides (MCT) and began treatment with UX007.
Groups:
- UX007: UX007 dosing was titrated to a target dose of 25-35% of total caloric intake or maximum tolerated dose. Participants were followed to evaluate the effects of UX007 over 24 weeks (Treatment Period), then continued treatment in the Extension Period for an additional 54 weeks for a total of 78 weeks of treatment.
Period: Overall Study
Arm/Group | UX007
Started | 29
Completed 24 Weeks of UX007 Treatment | 25
Completed | 24
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | UX007
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.06 (5.26)
Age, Customized [Count of Participants; unit: Participants]
  0 - 1 years | 2
  > 1 - 6 years | 13
  > 6 -18 years | 8
  > 18 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Time Adjusted-Area Under the Curve (AUC/Time) for Workload During Cycle Ergometry at Week 24
Description: To evaluate the impact 24 weeks of treatment with UX007 has on exercise intolerance, the change from Baseline in time adjusted-AUC (AUC/time) for workload during 40-minute cycle ergometry tests at Week 24 were assessed using the generalized estimation equation (GEE) model. A cycle ergometer can measure the work performed by an individual over time during physical exercise, the work was measured every 10 minutes from 0 to 40 minutes at Baseline and Week 24. The GEE model included the change from Baseline as the dependent variable, time as the categorical variable, and adjusted for Baseline measurement with compound symmetry covariance structure. An increase in AUC is reflective of improved exercise tolerance; a negative change from Baseline indicates worsening.
Time Frame: Baseline, Week 24
Population: Primary Analysis Set - Cycle Ergometry: the subset of participants in the primary analysis set (all enrolled participants who completed the 4 week Run-in Period and received at least one dose of UX007) who had at least one cycle ergometry test performed with any duration.
Measure: Least Squares Mean (Standard Error); unit: watts
Arm/Group | UX007
Number analyzed (Participants) | 7
watts | 423.594 (295.54)
Statistical Analysis 1: Comparison: UX007; Test type: Superiority; p = 0.1518, GEE model — The GEE model included the change from Baseline for each parameter as the dependent variable, time as the categorical variable, and adjusted for Baseline measurement with compound symmetry covariance structure; Least squares (LS) mean = 423.594, 95% CI 2-sided [-155.66 to 1002.85] — LS Mean, 95% confidence interval (CI), and p-values are based on the GEE model

2. Primary Outcome: Change From Baseline in Time-Adjusted-AUC for Respiratory Exchange Ratio (RER) During Cycle Ergometry at Week 24
Description: Change from baseline in time-adjusted-AUC for respiratory exchange ratio (RER) during cycle ergometry at Week 24, assessed using the GEE model, which included change from baseline as dependent variable, time as categorical variable, and adjusted for baseline measurement with compound symmetry covariance structure.
  RER during exercise is calculated as volume of carbon dioxide/volume of oxygen. RER measures whether carbohydrates or fats are being used as fuel. RER ≥1.0 indicates carbohydrates are the predominate fuel source. RER <1.0 and RER >0.70 indicates both fats and carbohydrates are the predominate fuel source. RER approximately =0.70 means fat is the predominant fuel source. RER would be expected to be lower, at similar exercise intensities, if a participant is able to utilize fat as an energy source. Therefore, an increase in RER (positive change from baseline) would suggest participants are still utilizing carbohydrates rather than fat, reflective a physiological response.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: respiratory exchange ratio
Arm/Group | UX007
Number analyzed (Participants) | 7
respiratory exchange ratio | -0.011 (0.0132)
Statistical Analysis 1: Comparison: UX007; Test type: Superiority; p = 0.3964, GEE model — [p-value comment as in outcome 1, analysis 1]; LS mean = -0.011, 95% CI 2-sided [-0.04 to 0.01] — LS Mean, 95% CI, and p-values are based on the GEE model

3. Primary Outcome: Change From Baseline in Actual Duration of Exercise During Cycle Ergometry at Week 24
Description: To evaluate the impact of 24 weeks of treatment with UX007 on exercise intolerance, the change from Baseline in actual duration of exercise during 40-minute cycle ergometry tests at Week 24 was assessed using the GEE model. The GEE model included the change from Baseline as the dependent variable, time as the categorical variable, and adjusted for Baseline measurement with compound symmetry covariance structure. Duration of exercise is expected to increase as exercise tolerance improves.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | UX007
Number analyzed (Participants) | 7
minutes | 4.671 (2.65)
Statistical Analysis 1: Comparison: UX007; Test type: Superiority; p = 0.0777, GEE model — [p-value comment as in outcome 1, analysis 1]; LS mean = 4.671, 95% CI 2-sided [-0.52 to 9.86] — LS Mean, 95% CI, and p-values are based on the GEE model

4. Primary Outcome: Change From Baseline in Distance Traveled During the 12-Minute Walk Test (12MWT) at Week 18
Description: To evaluate the impact 18 weeks of treatment with UX007 has on muscle function, the change from Baseline in distance traveled during a 12MWT at Week 18 was assessed using the GEE model. The GEE model included the change from Baseline as the dependent variable, time as the categorical variable, and adjusted for Baseline measurement with compound symmetry covariance structure. Distance traveled during the 12MWT is expected to increase as muscle function increases.
Time Frame: Baseline (last assessment during the 4-week run-in period), Week 18
Population: Primary Analysis Set - 12MWT: the subset of participants in the primary analysis set (all enrolled participants who completed the 4 week Run-in Period and received at least one dose of UX007) who had at least one 12MWT performed with any distance walked.
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | UX007
Number analyzed (Participants) | 8
meters | 181.37 (104.63)
Statistical Analysis 1: Comparison: UX007; Test type: Superiority; p = 0.0830, GEE model — [p-value comment as in outcome 1, analysis 1]; LS mean = 181.37, 95% CI 2-sided [-23.70 to 386.45] — LS Mean, 95% CI, and p-values are based on the GEE model

5. Primary Outcome: Change From Baseline in Energy Expenditure Index (EEI) During the 12MWT at Week 18
Description: To evaluate the impact 18 weeks of treatment with UX007 has on muscle function, the change from Baseline of EEI during the 12MWT at Week 18 was assessed using the GEE model. The GEE model included the change from Baseline as the dependent variable, time as the categorical variable, and adjusted for Baseline measurement with compound symmetry covariance structure. EEI is quantified as the post-test heart rate minus the pre-test heart rate (in beats/min) divided by overall velocity, and is valued in beats/meter. A decrease in EEI when walking a similar distance or no change when walking longer distances, may indicate improved exercise tolerance.
Time Frame: Baseline (last assessment during the 4-week run-in period), Week 18
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: beats/meter
Arm/Group | UX007
Number analyzed (Participants) | 8
beats/meter | -0.185 (0.09)
Statistical Analysis 1: Comparison: UX007; Test type: Superiority; p = 0.0320, GEE model — [p-value comment as in outcome 1, analysis 1]; LS mean = -0.185, 95% CI 2-sided [-0.35 to -0.02] — LS Mean, 95% CI, and p-values are based on the GEE model

6. Primary Outcome: Change From Baseline in Percentage of the Predicted 6-Minute Walk Test (6MWT) Distance Walked at Week 18
Description: To evaluate the impact 18 weeks of treatment with UX007 has on muscle function, the change from Baseline in the percentage of the predicted distance traveled during the first 6 minutes (6MWT) of the 12MWT at Week 18 was assessed using the GEE model. A participant's mathematical formula to calculate their percent predicted (PP) distance walked in the 6MWT was based on their demographics at baseline. For participants < 20 years old, the formula used was referenced from (Gieger, et. al. 2007) which calculated PP distance walked based on age, gender, and height. For participants >= 20 years old, the formula used was referenced from (Gibbons, et. al. 2001) and calculated the PP distance walked based on age and gender.
  The GEE model included the change from Baseline as the dependent variable, time as the categorical variable, and adjusted for Baseline measurement with compound symmetry covariance structure. Percent predicted values are expected to increase as muscle function increases.
Time Frame: Baseline (last assessment during the 4-week run-in period), Week 18
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: % of predicted distance (in meters)
Arm/Group | UX007
Number analyzed (Participants) | 8
% of predicted distance (in meters) | 12.44 (7.22)
Statistical Analysis 1: Comparison: UX007; Test type: Superiority; p = 0.0850, GEE model — [p-value comment as in outcome 1, analysis 1]; LS mean = 12.44, 95% CI 2-sided [-1.72 to 26.60] — LS Mean, 95% CI, and p-values are based on the GEE model

7. Primary Outcome: Change From Baseline in Physical Summary Score (PHS-10) of the Short Form 10 (SF-10) at Week 24
Description: To evaluate the impact treatment with UX007 has on functional disability and health in participants between 5 and 17 years of age, change from Baseline in the T-scores of the PHS-10 were assessed at Week 24 and analyzed using the GEE model. The GEE model included the change from Baseline as the dependent variable, time as the categorical variable, and adjusted for Baseline measurement with compound symmetry covariance structure.
  The SF-10 Health Survey for Children is a 10-item caregiver-completed assessment designed to measure children's health-related quality of life. The PHS-10 of the SF-10 is scored such that higher scores indicate more favorable functioning. The T-score based scoring signifies that scale scores are centered so that a score of 50 corresponds to the average score in a comprehensive sample of US population (scale scores are standardized to a mean of 50 and a standard deviation of 10).
Time Frame: Baseline, Week 24
Population: Primary Analysis Set - SF-10: the subset of participants in the primary analysis set (all enrolled participants who completed the 4 week Run-in Period and received at least one dose of UX007) who had at least one SF-10 test performed.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | UX007
Number analyzed (Participants) | 5
T-score | 2.16 (2.16)
Statistical Analysis 1: Comparison: UX007; Test type: Superiority; p = 0.3754, GEE model — The LS Mean, standard error (SE), 95% CI, and 2-sided p-value are from the GEE model; LS mean = 2.16, 95% CI 2-sided [-2.62 to 6.94]

8. Primary Outcome: Change From Baseline in Psychosocial Summary Score (PSS-10) of the SF10 at Week 24
Description: To evaluate the impact treatment with UX007 has on functional disability and health in participants between 5 and 17 years of age, changes from Baseline in the T-scores of the PSS-10 were assessed at Week 24 and analyzed using the GEE model. The GEE model included the change from Baseline as the dependent variable, time as the categorical variable, and adjusted for Baseline measurement with compound symmetry covariance structure.
  The PSS-10 of the SF-10 is scored such that higher scores indicate more favorable functioning. The T-score based scoring signifies that scale scores are centered so that a score of 50 corresponds to the average score in a comprehensive sample of US population (scale scores are standardized to a mean of 50 and a standard deviation of 10). Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values are indicative of more favorable functioning/better health.
Time Frame: Baseline, Week 24
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | UX007
Number analyzed (Participants) | 5
T-score | 0.816 (2.63)
Statistical Analysis 1: Comparison: UX007; Test type: Superiority; p = 0.7564, GEE model — The LS Mean, SE, 95% CI, and 2-sided p-value are from the GEE model; LS mean = 0.816, 95% CI 2-sided [-4.34 to 5.97]

9. Primary Outcome: Change From Baseline in the Physical Component Summary Scale (PCS-12) at Week 24
Description: Changes from baseline in T-scores as assessed by the PCS-12 Short-Form Health Survey, version 2 (SF-12v2) at Week 24 were assessed using the GEE model, which included the change from Baseline as the dependent variable, time as the categorical variable, and adjusted for Baseline measurement with compound symmetry covariance structure.
  PCS-12 scores were calculated from the individual responses to those questions that contribute to physical health. Raw scores range from 0 to 100 with higher scores indicating better health. The T-score based scoring signifies that scale scores are centered so that a score of 50 corresponds to the average score in the US general population (scale scores are standardized to a mean of 50 and a standard deviation of 10). Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values are indicative of more favorable functioning/better health.
Time Frame: Baseline, Week 24
Population: Primary Analysis Set - SF-12: the subset of participants in the primary analysis set (those who completed the 4-week run-in period and received at least one dose of UX007) who had at least one SF-12 test performed.
Measure: Least Squares Mean (Standard Deviation); unit: T-score
Arm/Group | UX007
Number analyzed (Participants) | 5
T-score | 8.88 (1.63)
Statistical Analysis 1: Comparison: UX007; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 1, analysis 1]; LS mean = 8.88, 95% CI 2-sided [5.67 to 12.08]

10. Primary Outcome: Change From Baseline in the Mental Component Summary Scale (MCS-12) at Week 24
Description: Changes from baseline of T-scores as assessed by the MCS-12 of the SF-12v2 at Week 24 were assessed using the GEE model, which included the change from Baseline as the dependent variable, time as the categorical variable, and adjusted for Baseline measurement with compound symmetry covariance structure.
  MCS-12 scores were calculated from the individual responses to those questions that contribute to mental health. Raw scores range from 0 to 100 with higher scores indicating better health. The T-score based scoring signifies that scale scores are centered so that a score of 50 corresponds to the average score in the US general population (scale scores are standardized to a mean of 50 and a standard deviation of 10). Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values are indicative of more favorable functioning/better health.
Time Frame: Baseline, Week 24
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | UX007
Number analyzed (Participants) | 5
T-score | 9.7 (4.0)
Statistical Analysis 1: Comparison: UX007; Test type: Superiority; p = 0.0152, GEE model — [p-value comment as in outcome 1, analysis 1]; LS mean = 9.70, 95% CI 2-sided [1.87 to 17.54] — LS Mean, 95% CI, and p-values are based on the GEE model

11. Primary Outcome: Annualized Event Rate of All Major Clinical Events Pre- and Post-Treatment With UX007
Description: Major clinical events are defined as adverse events (AEs) resulting in hospitalizations, emergency room (ER) visits, and emergency intervention.
Time Frame: 18 months before and after UX007 initiation
Population: Primary Analysis Set: participants who completed the 4-week run-in period and received at least one dose of UX007.
Measure: Mean (Standard Deviation); unit: events/year
Arm/Group | UX007
Number analyzed (Participants) | 29
events/year
  Pre-UX007 | 1.69 (1.6081)
  Post-UX007 | 0.877 (1.142)

12. Primary Outcome: Annualized Duration Rate of All Major Clinical Events Pre- and Post-Treatment With UX007
Description: Major clinical events are defined as AEs resulting in hospitalizations, ER visits, and emergency intervention.
Time Frame: 18 months before and after UX007 initiation
Population: Primary Analysis Set: participants who completed the 4-week run-in period and received at least one dose of UX007.
Measure: Mean (Standard Deviation); unit: days/year
Arm/Group | UX007
Number analyzed (Participants) | 29
days/year
  Pre-UX007 | 5.961 (6.0783)
  Post-UX007 | 2.964 (3.9733)

13. Primary Outcome: Annualized Event Rate of Major Rhabdomyolysis Clinical Events Pre- and Post-Treatment With UX007
Description: Rhabdomyolysis is a condition in which damaged skeletal muscle breaks down rapidly. Major rhabdomyolysis clinical events are defined as those AEs resulting in hospitalizations, ER visits, and emergency intervention.
Time Frame: 18 months before and after UX007 initiation
Population: Primary Analysis Set: participants who completed the 4-week run-in period and received at least one dose of UX007.
Measure: Mean (Standard Deviation); unit: events/year
Arm/Group | UX007
Number analyzed (Participants) | 29
events/year
  Pre-UX007 | 1.303 (1.5007)
  Post-UX007 | 0.833 (1.1513)

14. Primary Outcome: Annualized Duration Rate of Major Rhabdomyolysis Clinical Events Pre- and Post-Treatment With UX007
Description: as for outcome 13
Time Frame: 18 months before and after UX007 initiation
Population: Primary Analysis Set: participants who completed the 4-week run-in period and received at least one dose of UX007.
Measure: Mean (Standard Deviation); unit: days/year
Arm/Group | UX007
Number analyzed (Participants) | 29
days/year
  Pre-UX007 | 3.949 (4.3687)
  Post-UX007 | 2.792 (3.8452)

15. Primary Outcome: Annualized Event Rate of Major Hypoglycemia Clinical Events Pre- and Post-Treatment With UX007
Description: Major hypoglycemia clinical events are defined as those AEs resulting in hospitalizations, ER visits, and emergency intervention.
Time Frame: 18 months before and after UX007 initiation
Population: Primary Analysis Set: participants who completed the 4-week run-in period and received at least one dose of UX007.
Measure: Mean (Standard Deviation); unit: events/year
Arm/Group | UX007
Number analyzed (Participants) | 29
events/year
  Pre-UX007 | 0.318 (0.9053)
  Post-UX007 | 0.023 (0.1224)

16. Primary Outcome: Annualized Duration Rate of Major Hypoglycemia Clinical Events Pre- and Post-Treatment With UX007
Description: as for outcome 15
Time Frame: 18 months before and after UX007 initiation
Population: Primary Analysis Set: participants who completed the 4-week run-in period and received at least one dose of UX007.
Measure: Mean (Standard Deviation); unit: days/year
Arm/Group | UX007
Number analyzed (Participants) | 29
days/year
  Pre-UX007 | 1.414 (4.3025)
  Post-UX007 | 0.023 (0.1224)

17. Primary Outcome: Annualized Event Rate of Major Cardiac Clinical Events Pre- and Post-Treatment With UX007
Description: Major cardiac clinical events are defined as those AEs resulting in hospitalizations, ER visits, and emergency intervention.
Time Frame: 18 months before and after UX007 initiation
Population: Primary Analysis Set: participants who completed the 4-week run-in period and received at least one dose of UX007.
Measure: Mean (Standard Deviation); unit: events/year
Arm/Group | UX007
Number analyzed (Participants) | 29
events/year
  Pre-UX007 | 0.069 (0.2728)
  Post-UX007 | 0.021 (0.115)

18. Primary Outcome: Annualized Duration Rate of Major Cardiac Clinical Events Pre- and Post-Treatment With UX007
Description: as for outcome 17
Time Frame: 18 months before and after UX007 initiation
Population: Primary Analysis Set: participants who completed the 4-week run-in period and received at least one dose of UX007.
Measure: Mean (Standard Deviation); unit: days/year
Arm/Group | UX007
Number analyzed (Participants) | 29
days/year
  Pre-UX007 | 0.598 (2.4054)
  Post-UX007 | 0.149 (0.8047)

ADVERSE EVENTS:
Time Frame: From the first dose of UX007 through the Follow-up visit (Week 82) or 30 days following the last UX007 administration.
Description: Events presented are treatment-emergent. An event was considered as treatment-emergent if it occurred on or after the date of the first treatment of UX007.
Arm/Group | UX007
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 19/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UX007 (N=29)
Infection Prophylaxis (Surgical and medical procedures) | 1
Cardiomyopathy Acute (Cardiac disorders) | 1
Talipes (Congenital, familial and genetic disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Gastrointestinal Disorder (Gastrointestinal disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 11
Metabolic Disorder (Metabolism and nutrition disorders) | 1
Gastroenteritis (Infections and infestations) | 6
Gastroenteritis Viral (Infections and infestations) | 6
Gastrointestinal Viral Infection (Infections and infestations) | 2
Upper Respiratory Tract Infection (Infections and infestations) | 2
Adenoviral Upper Respiratory Infection (Infections and infestations) | 1
Adenovirus Infection (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Coxsackie Viral Infection (Infections and infestations) | 1
Croup Infectious (Infections and infestations) | 1
Otitis Media (Infections and infestations) | 1
Otitis Media Acute (Infections and infestations) | 1
Pneumonia Mycoplasmal (Infections and infestations) | 1
Respiratory Tract Infection Viral (Infections and infestations) | 1
Roseola (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UX007 (N=29)
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Pyrexia (General disorders) | 9
Pain (General disorders) | 3
Anxiety (Psychiatric disorders) | 2
Irritability (Psychiatric disorders) | 2
Panic Attack (Psychiatric disorders) | 2
Arthropod Bite (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 3
Laceration (Injury, poisoning and procedural complications) | 2
Procedural Pain (Injury, poisoning and procedural complications) | 2
Stoma Site Pain (Injury, poisoning and procedural complications) | 2
Blood Creatine Phosphokinase Increased (Investigations) | 3
Carnitine Decreased (Investigations) | 2
Tachycardia (Cardiac disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 2
Headache (Nervous system disorders) | 9
Eye Swelling (Eye disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 13
Abdominal Pain (Gastrointestinal disorders) | 8
Abdominal Pain Upper (Gastrointestinal disorders) | 4
Gastrointestinal Pain (Gastrointestinal disorders) | 3
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3
Abdominal Distension (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Teething (Gastrointestinal disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 3
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2
Decreased Appetite (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 2
Upper Respiratory Tract Infection (Infections and infestations) | 11
Ear Infection (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 5
Bronchitis (Infections and infestations) | 4
Gastroenteritis Viral (Infections and infestations) | 4
Gastrointestinal Viral Infection (Infections and infestations) | 4
Rhinitis (Infections and infestations) | 4
Viral Upper Respiratory Tract Infection (Infections and infestations) | 4
Conjunctivitis (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 3
Urinary Tract Infection (Infections and infestations) | 3
Otitis Media (Infections and infestations) | 2
Respiratory Tract Infection Viral (Infections and infestations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.